CLINICAL TRIAL: NCT04521673
Title: Pathogen Detection in Infectious Uveitis in China
Brief Title: Pathogen Detection in Infectious Uveitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ping Fei, Associate professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-20-014
Record Dates: First submitted 2020-08-19; First posted 2020-08-20 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Infectious Panuveitis; Infectious Iridocyclitis
Keywords: infectious uveitis; pathogen; PCR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Aqueous Humor and vitreous
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- infectious uveitis: Patients suffering from suspected infectious uveitis, who have vitrectomy performed for diagnostic purpose or anterior chamber tap
- Control group: Patients suffering from either cataract surgery or vitrectomy who has been ruled out for infectious ocular diseases

SUMMARY:
Infectious uveitis is a very important blinding disease. Some people who have been diagnosed with idiopathic uveitis may also have the activity of pathogens in the eye. However, due to the limitation of the amount of ocular samples, it is difficult to make a rapid and effective diagnosis of infection.Current study is to explore the infective cause of uveitis in China by using a broad diagnostic approach of detection.

DETAILED DESCRIPTION:
Infectious uveitis is a very important blinding disease. Some people who have been diagnosed with idiopathic uveitis may also have the activity of pathogens in the eye. However, due to the limitation of the amount of ocular samples, it is difficult to make a rapid and effective diagnosis of infection.

The study is to explore the infective cause of uveitis in China by using a broad diagnostic approach of detection, including multiple molecular bio-techniques. We also plan to explore the distribution of pathogens in infectious uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient at a referal hospital eye clinic with clinically suspected infectious uveitis

Exclusion Criteria:

* Patients not eligible for the Inclusion Criteria
* Confirmed auto-immune uveitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patient at a referal hospital eye clinic with clinically suspected infectious uveitis, who undergo AC tap or diagnostic vitrectomy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence and distribution of intraocular infections in the study group | Oct 2020 to Sep 2022
  Prevalence and distribution of intraocular infections in the study group

SECONDARY OUTCOMES:
The sensitivity and specificity of multiple molecular diagnostic methods for detection of bacteria or virus fungi in the study group | Oct 2020 to Sep 2022
  The sensitivity and specificity of multiple molecular diagnostic methods for detection of bacteria or virus fungi in the study group

CONTACTS AND LOCATIONS:
Overall Officials: Ping Fei, MD，PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 2 years after the study
Access Criteria: if required propriately